CLINICAL TRIAL: NCT05692596
Title: The Pancreas Interception Center (PIC) for Early Detection, Prevention, and Novel Therapeutics
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22156
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cyst; Chronic Pancreatitis; Fatty Pancreas; Genetic Pancreatic Cancer; Genetic Pancreatitis; BRCA Mutation; Lynch Syndrome; FAP; Familial Atypical Multiple Mole-Melanoma; PALB2 Gene Mutation; Peutz-Jeghers Syndrome; Ataxia Telangiectasia
Keywords: pancreas; database
MeSH Terms: conditions — Pancreatic Cyst; Pancreatitis, Chronic; Colorectal Neoplasms, Hereditary Nonpolyposis; Dysplastic Nevus Syndrome; Peutz-Jeghers Syndrome; Ataxia Telangiectasia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Participants include patients scheduled to see the clinical team in the Pancreas Interception Center (PIC) which will be housed in the Moffitt GI Clinic.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Investigators will compile data typically collected clinically. This data will include demographics, cancer screening procedures, cancer diagnosis and staging, chemotherapy, immunotherapy, radiation therapy, surgery, comorbidities, medication use, lifestyle and other cancer risk factors, quality of life, vital status, and molecular data generated from specimens collected clinically.

SUMMARY:
The long-term goal of our PIC is to develop effective strategies that can be applied clinically at the point-of-care to prevent, intercept, or detect PDAC at an early stage, thereby reducing PDAC burden and saving lives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Moffitt Cancer Center patients presenting with a pancreatic cyst, and/or inherited syndrome that predisposes them to pancreatic ductal adenocarcinoma (PDAC)
* Moffitt Cancer Center patients undergoing evaluation for localized/early stage PDAC.
* Moffitt Cancer Center patients with a combination of PDAC risk factors such as a history of chronic or new-onset diabetes, pancreatitis, obesity, tobacco exposure, toxin exposure and/or heavy alcohol consumption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the Moffitt GI clinic
Sampling Method: Non-Probability Sample
Enrollment: 317 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Database creation | 24 months
  A centralized, real-time, queryable and secure database will be developed that will integrate data on Moffitt patients diagnosed with pancreatic ductal adenocarcinoma (PDAC), pancreatic cystic lesions (benign, pre-cancerous and malignant), or an inherited PDAC susceptibility.

CONTACTS AND LOCATIONS:
Overall Officials: Shaffer Mok, MD, MBS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided